CLINICAL TRIAL: NCT02399553
Title: Effect of the Interaction Between the Type of Artificial Turf and Boots Model of Bone Health in Children Soccer Players
Acronym: FUTBOMAS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad de Zaragoza (Other)
Responsible Party: Principal Investigator, José A. Casajús, Proffesor, Universidad de Zaragoza
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: DEP 2103-32724
Record Dates: First submitted 2015-03-20; First posted 2015-03-26 (Estimated); Last update posted 2016-05-12 (Estimated); Status verified 2016-05

CONDITIONS: Soccer; Bone Density; Physical Fitness

ARMS (5):
- Soccer 2G (Experimental): Soccer players who trained in second generation artificial turf
  Interventions: Other: Soccer boot intervention
- Soccer 3G (Experimental): Soccer players who trained in third generation artificial turf
  Interventions: Other: Soccer boot intervention
- Soccer NG (Experimental): Soccer players who trained in natural grass
  Interventions: Other: Soccer boot intervention
- Soccer NON-NG (Experimental): Soccer players who trained in non-natural grass
  Interventions: Other: Soccer boot intervention
- Control group (No Intervention)

INTERVENTIONS:
Other: Soccer boot intervention
  Arms: Soccer 2G; Soccer 3G; Soccer NG; Soccer NON-NG

SUMMARY:
The number of turf fields has experienced an important increase in public and private facilities during the last years. This artificial surface will be predominant in any soccer field in the next years. Among turf fields there are many different types depending on their construction characteristics (with and without asphalted base, elastic base, rubber filling, etc.). Officially all types of artificial turfs should have similar stability and impact absorption characteristics. On the other hand there is a great variety of soccer-boots, especially for youth soccer players, similar to the football stars.

Many evidences support the fact that when a person exercises many different type of impacts-stimulus are necessary in order to stimulate bone and skeletal muscle systems. However, it is not known yet whether this effect can be extended or shortened depending on the type of artificial surface and soccer-boots used, or even more whether it could be more or less dangerous and/or provoke injuries/disagreement among the users. Little information is available in youth soccer player pointing in the same direction but still controversial. Furthermore, bone strength do not only depends on bone mass but on bone structure and microarchitecture. The cross sectional area, cortex thickness or trabecular density are important aspects of bone health. There are few studies on the effect of interaction between turf field and soccer boots on bone architecture of youth soccer players. This information is relevant for present and future health of adolescents practicing football and for all the organizations promoting this sport.

Due to the fact that turf fields are preferentially used by youth populations, it is important to know the real effects of the interaction between of different type of artificial surfaces and soccer boots on children bone mass development. Nowadays, there are no data and/or defined guidelines that can answer those unresolved questions, thus the main aim of the present project is to identify which turf field and soccer boots are the most adequate to optimize the acquisitions of bone mass in children soccer players.

ELIGIBILITY:
Inclusion Criteria:

* Both: Aged from 11-13 years.
* Both: Parental/guardian permission (informed consent) and if appropriate, child verbal assent.
* Specific for the control group: Subjects that do not perform more than 3 hours of physical activity per week.

Exclusion Criteria:

* Taking medication affecting bone.
* Non-Caucasian.

Ages: 11 Years to 13 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 129 (Actual)
Dates: Start 2013-09; Primary Completion 2016-01 (Actual); Study Completion 2016-01 (Actual)

PRIMARY OUTCOMES:
Change in body composition during 2 years evaluated by Dual energy X-ray absorptiometry | Change from baseline in body composition at 2 years

CONTACTS AND LOCATIONS:
Locations (1):
- José Antonio Casajús Mallén, Zaragoza, Zaragoza, Spain